CLINICAL TRIAL: NCT07107399
Title: Therapeutic Effect of Microfragmented Adipose Tissue (Lipogems) Injection on Maximum Interincisal Opening Versus Injectable Platelet-rich Plasma (PRP) for the Treatment of Anterior Disc Displacement With Reduction : A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed hosni, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tmj injection
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: TMJ Disc Disorder
Keywords: lipogem

STUDY DESIGN:
Intervention Model Description: B) Injectable Lipogems, a form of adipose (fat) tissue-derived regenerative medicine, is an emerging treatment for a variety of musculoskeletal conditions, including TMJ disorders such as anterior disc displacement with reduction. Lipogems involves harvesting and processing a small amount of the patient's own fat tissue, then injecting it into the affected area. Here's why Lipogems is considered an important option in treating TMJ disorders with anterior disc displacement with reduction.
  Lipogems contains a rich concentration of regenerative cells, such as mesenchymal stem cells (MSCs), along with growth factors, cytokines, and other bioactive molecules. These components play a crucial role in tissue regeneration, healing, and the repair of damaged structures within the TMJ, such as the articular disc, ligaments, and surrounding tissues. These growth factors can support the healing process of the damaged tissues that may be contributing to the disc displacement.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet-rich plasma (Active Comparator)
  Interventions: Other: platelet-rich plasma
- microfragmented adipose tissue (Experimental)
  Interventions: Other: microfragmented adipose tissue

INTERVENTIONS:
Other: microfragmented adipose tissue — Receive micro fragmented adipose tissue obtained from the buccal pad of fat after arthrocentessis.
  * Direct access to the buccal fat pad, is found at distobuccal depth of the maxillary tuberosity.
  * It may be dissected during the resection an upper mucosal incision posterior to the second molar
  * After a single scissor stab through the periosteum the (BFP)extrude into the operative site.
  * Closure of the flap by suitable suture.
  * Collection of lipids then manually manipulated with two syringes connecting together and pushing the lipids against each other to receive the injectable amount of micro fragmented adipose tissue .
  * Ready for TMJ injection.
  Arms: microfragmented adipose tissue
Other: platelet-rich plasma — I - double-puncture arthrocentesis technique was followed, and 300 mL of Ringer's lactate solution was used to irrigate the joint space through the marked points . After arthrocentesis PRP was prepared from 5 mL of autologous venous blood sample taken from the antecubital vein. The collected blood was then transferred to a test tube containing 0.5 mL of sodium citrate (anticoagulant) (0.5 mL) and was centrifuged at a rate of 2100 rpm for 15 min. The plasma from the first harvest was fractionated by centrifugation at 3500 rpm for 10 min to prepare PRP.
  Arms: platelet-rich plasma

SUMMARY:
this procedure is to remove inflammatory mediators, reduce friction, stimulate the production of new synovial fluid, eliminate suction-cup effect.

The purpose of this study was to evaluate the hypothesis that TMJ arthrocentesis with injection of autologous micro fragmented adipose tissue leads to better clinical outcomes in terms of reducing pain and improving function compared with arthrocentesis and injection of platelets rich plasma (prp)in patients with TMJ internal derangement and osteoarthritis.

Preliminary results of this clinical trial show that the injection of micro fragmented adipose tissue can significantly improve outcomes of pain and function compared with the standard treatment and encourage to pursue research on this topic.

Further studies with a longer follow-up time are needed to evaluate the clinical stability of the achieved improvement in pain and function.

For this reason, this protocol has been designed with the aim to investigate whether injection in the TMJ of micro fragmented fat tissue can achieve the same improvements of pain and function, compare this technique with prp injection.

DETAILED DESCRIPTION:
Anterior disc displacement with reduction (DDwR) of the temporomandibular joint (TMJ) is a prevalent condition characterized by the displacement of the articular disc during jaw movement, often leading to pain, clicking sounds, and restricted mouth opening. Traditional treatments include conservative approaches such as physical therapy, occlusal splints, and pharmacological interventions. However, for patients unresponsive to these methods, intra-articular injections of regenerative therapies like microfragmented adipose tissue (MFAT) and platelet-rich plasma (PRP) have emerged as promising alternatives.

Arthrocentesis first described by Nitzan et al. [1.2] is the simplest intervention on the TMJ with the aim to decrease joint pain and improve the range of motion in patients not responding to initial conservative treatment.

Arthrocentesis consists of an intraarticular lavage using 2 needles placed in the upper joint space. It is a versatile technique which can be performed under local anesthesia in an outpatient setting as well Arthrocentesis has been demonstrated to be a very effective procedure with a high success rate and a favorable benefit-cost ratio.

In addition to arthrocentesis:

Microfragmented Adipose Tissue (MFAT) Injections MFAT involves the extraction and processing of adipose tissue to create a suspension rich in mesenchymal stem cells, growth factors, and extracellular matrix components. This suspension is then injected into the affected joint to promote tissue repair and reduce inflammation.

A study published in Stem Cells Translational Medicine in 2023 evaluated the efficacy of MFAT injections in patients with knee osteoarthritis. The results demonstrated significant improvements in joint pain and functionality, with median changes in the Knee injury and Osteoarthritis Outcome Score (KOOS) Pain subscale ranging from 18.1 at week 2 to 27.8 at 1 year. These findings suggest that MFAT may be a viable alternative treatment for patients with joint conditions who fall into the orthopedic treatment gap.

While this study focused on knee osteoarthritis, the regenerative properties of MFAT suggest potential applicability to TMJ disorders. However, further research is needed to confirm its effectiveness in the TMJ context.

Platelet-Rich Plasma (PRP) Injections PRP therapy involves concentrating platelets from the patient's own blood and injecting them into the affected joint to stimulate healing.

A systematic review published in BMC Oral Health in 2024 examined the effectiveness of PRP injections for TMJ disorders. The review concluded that PRP injections, particularly when combined with arthrocentesis, were effective in reducing pain and improving mandibular function in patients with TMJ internal derangement.

Additionally, a study in the Open Journal of Stomatology in 2023 evaluated the effect of platelet-rich growth factors (PRGFs) in the treatment of TMJ disc displacement. The results indicated that PRGFs could be a possible alternative treatment for patients who did not respond to standard treatments, showing early efficacy in reducing pain and improving joint function.

Comparative Efficacy While both MFAT and PRP injections have demonstrated efficacy in treating joint disorders, direct comparative studies in the context of TMJ anterior disc displacement with reduction are limited. The existing literature primarily focuses on individual therapies rather than head-to-head comparisons. Therefore, it is challenging to definitively conclude which treatment offers superior outcomes for TMJ disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have one or more signs and symptoms of these

  * Disc displacement assessed by clinical examination and MRI
  * Symptoms: Patients who report typical symptoms of TMJ dysfunction, such as pain, discomfort, or clicking sounds in the joint, especially when opening or closing the mouth.
  * Mouth Opening: Limited range of motion or difficulty with full mouth opening .
  * Clicking: Audible clicking.
  * Pain: Pain or tenderness around the TMJ, often radiating to the ear, temple, or neck.

Exclusion Criteria:

* Previously diagnosed hematological and neurological conditions;

  * Previous malignant head and neck neoplasms;
  * Contraindication to fat harvesting.
  * Uncooperative patients.
  * connective tissue disorders.
  * a pacemaker or any other metal prosthesis in the body.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
maximum interincisal opening | 1 week , 3 months
  maximum interincisal opening and it is measured by caliper in mm

SECONDARY OUTCOMES:
change in pain severity | 1 week , 3 months
  pain severity will be assessed using vas scale (0-10) where 0 = no pain and 10 = sever pain . participants will report their pain level at each time point
presence or absence of joint clicking (binary outcome) | 1 week , 3 months
  joint clicking will be assessed as a binary outcome (yes/no)based on the clinical examination and patient-reported symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hosni Ahmed Hosni Ali, bachelor's degree, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mittal A, Klarie SJ, Sharma S, Roy B, Paul JI, Sharma S. Efficacy of Intra-articular Platelet-rich Plasma versus Hydrocortisone with Local Anaesthetic Injection in Temporomandibular Joint Disorders - A Prospective Study. Ann Maxillofac Surg. 2024 Jul-Dec;14(2):166-170. doi: 10.4103/ams.ams_237_23. Epub 2024 Sep 11. PMID 39957867